CLINICAL TRIAL: NCT05906043
Title: A Multidisciplinary Approach to Assessing and Treating Fatigue in Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Dublin (Other)
Responsible Party: Principal Investigator, Hugh Mulcahy, Prof. Hugh Mulcahy, FRCPI MD, University College Dublin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RS22-038
Record Dates: First submitted 2023-05-24; First posted 2023-06-15 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Inflammatory Bowel Diseases; Fatigue
MeSH Terms: conditions — Inflammatory Bowel Diseases; Fatigue | interventions — Acceptance and Commitment Therapy; Probiotics

STUDY DESIGN:
Intervention Model Description: Cross sectional study, with observational elements and four interventions utilising a single case experimental design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cross Sectional Study to define the extent and severity of fatigue (No Intervention): All patients attending the IBD service that meet inclusion criteria will be given the opportunity to participate in this study. Information will be collected at baseline including demographic data, IBD history and symptoms, co-morbidities and disease activity. Patients will have baseline blood tests taken to assess for causes of fatigue as well as faecal calprotectin to assess for evidence of inflammation. Patients without fatigue will at this point exit the study and will not require any further follow up.
- Treatment for active disease and its effect on fatigue. (No Intervention): A longitudinal study of contemporary treatment for active disease and its effect on fatigue. Patients with active disease and fatigue will be followed prospectively while undergoing treatment for active IBD with the IBD team. If their fatigue resolves, they will exit the study at this point. If their fatigue persists, they will be further assessed as detailed below.
- The effect of treating anaemia on fatigue in IBD (No Intervention): A longitudinal study assessing anaemia and the effect of treatment on fatigue in those subjects with inactive IBD.Patients with anaemia and fatigue will be followed prospectively while undergoing treatment for anaemia with the IBD team. The study outcomes will be assessed at recruitment and when their anaemia has resolved (this may occur in parallel with the disease activity arm). If their fatigue resolves, they will exit the study at this point. If their fatigue persists, they will be further assessed as detailed below.
- Assessing exercise therapies in IBD subjects with fatigue (Other): A longitudinal study assessing of dietary and exercise therapies for IBD subjects with fatigue using a single case study (SCS) design. They will have their physical activity levels assessed at recruitment and as needed after active disease/anaemia/nutritional deficiencies have been adequately treated. Those with fatigue despite optimisation will be offered a physical activity intervention. Each participant will be assessed initially and subsequently assigned a physical activity intervention with a physical therapist.
  Interventions: Behavioral: Exercise Intervention
- Acceptance and commitment therapy (ACT) in IBD subjects with fatigue (Other): A longitudinal study of acceptance and commitment therapy (ACT) in IBD subjects with psychological disability and fatigue using a single case study (SCS) design. All patients will undergo psychological assessment as detailed above at recruitment and as needed after active disease/anaemia/nutritional deficiencies have been adequately treated. Those with fatigue and psychological disability will be referred to the IBD psychology service or recruited to a psychological intervention. Participants will receive an online intervention with a psychologist from the School of Psychology in University College Dublin to address psychological disability and associated fatigue.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- ACT for IBD subjects with sleep disturbance and fatigue (Other): A longitudinal study of ACT for IBD subjects with sleep disturbance using a single case study (SCS) design. Patients will have their sleep quality assessed at recruitment and as needed after active disease/anaemia/nutritional deficiencies have been adequately treated. Those with sleep disturbance will undergo sleep studies at home both at the start and end of the intervention. This device will be a non-invasive, widely available sleep device worn on the wrist or the patient's index finger for one to three consecutive nights. They will be referred to the sleep medicine unit in SVUH if sleep apnea or another diagnosis that requires medical intervention is identified. Otherwise they will undergo an online intervention with a psychologist from the School of Psychology in University College Dublin to address their sleep quality.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- A longitudinal study of probiotics for IBD subjects with fatigue (Other): Participants will have their stool analysed to assess the diversity of their microbiome. They will receive a twelve-week course of a probiotic which will be taken once daily. They will then have their stool re-assessed at the completion of the intervention.
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Behavioral: Exercise Intervention — Exercise intervention
  Arms: Assessing exercise therapies in IBD subjects with fatigue
Behavioral: Acceptance and Commitment Therapy — ACT will be used for patients with psychological disability as well as for those with sleep disturbance
  Arms: ACT for IBD subjects with sleep disturbance and fatigue; Acceptance and commitment therapy (ACT) in IBD subjects with fatigue
Dietary Supplement: Probiotic — Use of a probiotic
  Arms: A longitudinal study of probiotics for IBD subjects with fatigue

SUMMARY:
This study is examining fatigue in patients with Inflammatory Bowel Disease (IBD). IBD includes Ulcerative Colitis (UC) and Crohn's disease. These are inflammatory conditions of the gastrointestinal tract and are associated with symptoms including diarrhoea, rectal bleeding and abdominal pain. Fatigue is a common problem for patents with IBD, affecting 80% of patients with active disease.This study aims to identify all IBD patients with fatigue. Initially, the investigators will address all medical causes of fatigue in line with current practice, using a stepwise approach (e.g. assessing for and treating active inflammation, anaemia as well as electrolyte, hormone and vitamin imbalances). The aim is to treat fatigue using a detailed algorithm, as fatigue is often a consequence of multiple issues in IBD patients. The investigators will assess the role of physical activity, nutritional status and psychological wellbeing in fatigue persisting in medically-optimised IBD patients. In addition, the contribution of the microbiome to fatigue will be assessed. For those in whom these factors are identified alongside persistent fatigue, interventions have been designed to address these factors and the resulting fatigue.

DETAILED DESCRIPTION:
This is a longitudinal research study to define the extent and severity of fatigue in IBD patients; patients will be followed for a period of weeks to months depending on each individual participants needs. The study will be a cross-sectional in nature initially. The study is open to all mobile and non-pregnant Crohn's disease and ulcerative colitis patients between the ages of 18 and 70 years. Recruitment will take place in St Vincent's University Hospital, an academic teaching hospital, from Gastroenterology clinics as well as through the IBD clinical nurse specialist service. Patients that meet inclusion criteria will be recruited from clinics and/or through the IBD clinical nurse specialist service. The recruited subjects will be briefed on the inclusion and exclusion criteria, the nature of the study as well as the outcome measure. Participants will receive information packs and consent forms. All participants will have the opportunity to withdraw at any stage during the study and this will be explained to them. Patients will be followed up as clinically necessary within the parameters of the study and at the IBD clinic at clinically appropriate intervals. All patients attending the IBD service that meet inclusion criteria will be given the opportunity to participate in this study. Information will be collected at baseline including demographic data, IBD history and symptoms, co-morbidities and disease activity.

There are seven elements to this study that will be carried out in parallel:

1. An initial cross-sectional study to define the extent and severity of fatigue in IBD subjects incorporating a simple fitness test protocol. All patients attending the IBD service that meet inclusion criteria will be given the opportunity to participate in this study. Information will be collected at baseline including demographic data, IBD history and symptoms, co-morbidities and disease activity. Patients will have baseline blood tests taken to assess for causes of fatigue as well as faecal calprotectin to assess for evidence of inflammation. Patients without fatigue will at this point exit the study and will not require any further follow up. In those with fatigue, disease activity will be assessed and treated in accordance with current clinical guidelines (as would be standard of care). Fatigued patients will also be assessed for anaemia and other medical causes of fatigue and treated for these as per current clinical practice guidelines.
2. A longitudinal study of contemporary treatment for active disease and its effect on fatigue. Patients with active disease and fatigue will be followed prospectively while undergoing treatment for active IBD with the IBD team. Each patient's response to treatment will vary and so the exact time point between disease treatment and resolution of disease activity cannot be clearly defined. The study outcomes will be assessed at recruitment and when participants achieve clinical and biochemical remission. If fatigue resolves, participants will exit the study at this point. If fatigue persists, further assessments will take place as detailed below.
3. A longitudinal study assessing anaemia and the effect of treatment on fatigue in those subjects with inactive IBD. Patients with anaemia and fatigue will be followed prospectively while undergoing treatment for anaemia with the IBD team. Each patient's response to treatment will vary and so the exact time point between anaemia treatment and resolution of anaemia cannot be clearly defined. The study outcomes will be assessed at recruitment and when anaemia has resolved (this may occur in parallel with the disease activity arm). If fatigue resolves, participants will exit the study at this point. If fatigue persists, further assessments will take place as detailed below.
4. A longitudinal study assessing of dietary and exercise therapies for IBD subjects using a single case study (SCS) design. Participants will also have physical activity levels assessed at recruitment and as needed after active disease/anaemia/nutritional deficiencies have been adequately treated. These assessments will take place on site in St Vincent's University Hospital. If fatigue resolves, participants will exit the study at this point. Those with fatigue despite optimizing nutrition will be offered a physical activity intervention. The time interval between recruitment and resolution of micronutrient deficiencies will vary from patient to patient and so the exact time interval cannot be specified. Each participant will be assessed initially and subsequently assigned a physical activity intervention with a physical therapist designed by the Department of Sports Medicine, University College Dublin.
5. A longitudinal study of acceptance and commitment therapy (ACT) in IBD subjects with psychological disability using a single case study (SCS) design. All patients will undergo psychological assessment as detailed above at recruitment and as needed after active disease/anaemia/nutritional deficiencies have been adequately treated. Those with fatigue and psychological disability will be referred to the IBD psychology service or recruited to a psychological intervention. Participants will receive an intervention with a psychologist from the School of Psychology in University College Dublin to address psychological disability and associated fatigue.
6. A longitudinal study of ACT for IBD subjects with sleep disturbance using a single case study (SCS) design. Patients will have sleep quality assessed at recruitment and as needed after active disease/anaemia/nutritional deficiencies have been adequately treated. Those with sleep disturbance will undergo sleep studies at home both at the start and end of the intervention. This device will be a non-invasive, widely available sleep device worn on the wrist or the patient's index finger for one to three consecutive nights. Participants will be referred to the sleep medicine unit in SVUH if sleep apnea or another diagnosis that requires medical intervention is identified. Otherwise participants will undergo an intervention with a psychologist from the School of Psychology in University College Dublin to address sleep quality.
7. A longitudinal study of probiotics for IBD subjects with fatigue. Participants will have stool samples analysed to assess the microbiome diversity. A twelve-week course of a probiotic which will be taken once daily will then be provided. Stool will be re-assessed at the completion of the intervention.

Each of the four treatment arms will be treated as multiple baseline single case experimental design (SCED). Thus, each participant is treated as an individual study. This type of study provides evidence for the effectiveness of interventions with much fewer participants than group average-based designs such as Randomized Controlled Trials. Standard group-based designs may find an overall treatment benefit on average but may underestimate risks, ineffectiveness, and benefits to the individual.

Each participant will receive a follow up phone call after the intervention is complete, to identify any challenges integrating skills discussed during the interventions. Completion of an online questionnaire will be required at the end of the study period, in order to assess the primary and secondary outcomes.

Any participants with ongoing fatigue will be able to opt to participate in the remaining treatment arms if needed.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of inflammatory bowel disease

Exclusion Criteria:

* Pregnant women
* Patients unable to consent
* Patients under 18 and over 70 years of age

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-06-24 (Estimated); Study Completion 2025-08-24 (Estimated)

PRIMARY OUTCOMES:
Fatigue | Dependent on the factors involved; this will be different for each participant (up to 24 months)
  The primary outcome is to assess for improvement in fatigue using the Multidimensional Fatigue Index (MFI). This is a 20 item scale; each item is scored 1 to 5 with higher scores indicating higher levels of fatigue. Total score for each participant will range between 20 and 100; with high scores indicating more fatigue.

SECONDARY OUTCOMES:
Physical activity | Intervention will take place over 12 weeks
  Assessing changes in activity based on the International Physical Activity Questionnaire (IPAQ). The sum score is expressed in physical activity Metabolic Equivalent of Task (MET)-minutes per day or week. Higher scores indicate higher levels of activity.
Work Productivity and Activity Impairment | Intervention will take place over 12 weeks
  Assessing changes in Work Productivity and Activity Impairment Questionnaire (WPAIQ). The score for the WPAIQ is expressed as a percentage. Higher percentages of work and activity impairment indicating worse outcomes.
Physical activity: Grip strength | Intervention will take place over 12 weeks
  Assessing changes in grip strength. This is measured in kilograms. Higher grip strength in kilograms indicate better outcomes (values are age dependent).
Physical activity: Power assessment | Intervention will take place over 12 weeks
  Assessing changes in squat testing: Time taken for 5 squats in seconds assesses power. The shorter the time, the higher the power.
Physical activity: endurance assessment | Intervention will take place over 12 weeks
  Assessing changes in squat testing. The thirty-second sit to stand test will assess endurance. The higher the number of squats performed suggests higher levels of endurance and leg strength.
Physical activity: weight | Intervention will take place over 12 weeks
  Assessing changes in weight using bioimpedance analysis as part of the physical assessment. This will be measured in kilograms.
Psychological assessment | Intervention will take place over 12 weeks
  Depression, Anxiety and Stress Scale (DASS-21) will be used. Participants will score between 0-63 with higher scores indicating worse outcomes and increased anxiety, depression and stress levels.
Personality assessment | Intervention will take place over 12 weeks
  The Big Five Personality Inventory. This measures personality traits using 10 questions measured on a 5 point scale. This is to assess the impact of personality traits on fatigue rather than correlating directly with better or worse outcomes.
Disease related disability and quality of life | Dependent on the factors involved; this will be different for each participant (up to 24 months)
  IBD Disability index. Scores range from 0-100. Higher scores indicate worse outcomes.
Health related quality of life | Dependent on the factors involved; this will be different for each participant (up to 24 months)
  Short Health Scale (SHS) is a four part visual analogue scale questionnaire; the scale is marked from 0 to 100mm. Higher scores indicate a negative impact of disease on quality of life.
Sleep quality | Intervention will take place over 12 weeks
  Epworth Sleepiness Scale is scored from 0 to 24 with scores above 12 indicating abnormal levels of daytime somnolence.
Body image | Dependent on the factors involved; this will be different for each participant (up to 24 months)
  Modified Body Image Scale. This scale includes nine items scored 0 to 3. Score ranges from 0 to 27 with higher scores indicating increased body image dissatisfaction.
Nutritional assessment | Dependent on the factors involved; this will be different for each participant (up to 24 months)
  Malnutrition Universal Screening Tool (MUST). There are three measurements assessed; total score ranges from 0 to 6 with a score above 2 indicating worse outcomes.
Disease activity for participants with Ulcerative Colitis | Dependent on the factors involved; this will be different for each participant (up to 24 months)
  Partial Mayo score for patients with Ulcerative Colitis (See outcome 16 for the applicable scoring system from participants with Crohns disease). Parameters of disease activity are scored 0 to 3 with a total score range of 0 to 9. Higher scores correlate with higher levels of disease activity.
Disease activity for participants with Crohn's disease | Dependent on the factors involved; this will be different for each participant (up to 24 months)
  Crohns disease activity index score ranges from 0 to 600. A score of less than 150 indicates disease in remission. Higher scores correlate with higher levels of disease activity.
C-Reactive Protein Concentration: Serum marker of inflammation to assess disease activity | Dependent on the factors involved; this will be different for each participant (up to 24 months)
  CRP is a serum measurement of inflammation. Normal range is 0-5mg/L. Higher values indicate higher levels of systemic inflammation.
Faecal calprotectin concentration: Stool analysis to assess for disease activity | Dependent on the factors involved; this will be different for each participant (up to 24 months)
  Faecal calprotectin. This is a measure of disease activity. Values less than 250 micrograms/miligrams indicate disease remission. Higher values indicate disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Mulcahy, MD FRCPI, Principal Investigator — St Vincent's University Hospital, Ireland
Locations (1):
- St Vincent's University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will be anonymised in accordance with EU Data Protection legislation. Anonymised data will be available upon request.

REFERENCES:
- [Background] Villoria A, Garcia V, Dosal A, Moreno L, Montserrat A, Figuerola A, Horta D, Calvet X, Ramirez-Lazaro MJ. Fatigue in out-patients with inflammatory bowel disease: Prevalence and predictive factors. PLoS One. 2017 Jul 27;12(7):e0181435. doi: 10.1371/journal.pone.0181435. eCollection 2017. PMID 28749985
- [Background] Minderhoud IM, Samsom M, Oldenburg B. Crohn's disease, fatigue, and infliximab: is there a role for cytokines in the pathogenesis of fatigue? World J Gastroenterol. 2007 Apr 14;13(14):2089-93. doi: 10.3748/wjg.v13.i14.2089. PMID 17465453
- [Background] van Langenberg DR, Gibson PR. Systematic review: fatigue in inflammatory bowel disease. Aliment Pharmacol Ther. 2010 Jul;32(2):131-43. doi: 10.1111/j.1365-2036.2010.04347.x. Epub 2010 May 6. PMID 20456309
- [Background] Jelsness-Jorgensen LP, Bernklev T, Henriksen M, Torp R, Moum BA. Chronic fatigue is more prevalent in patients with inflammatory bowel disease than in healthy controls. Inflamm Bowel Dis. 2011 Jul;17(7):1564-72. doi: 10.1002/ibd.21530. Epub 2010 Nov 8. PMID 21674713
- [Background] Grimstad T, Norheim KB, Isaksen K, Leitao K, Hetta AK, Carlsen A, Karlsen LN, Skoie IM, Goransson L, Harboe E, Aabakken L, Omdal R. Fatigue in Newly Diagnosed Inflammatory Bowel Disease. J Crohns Colitis. 2015 Sep;9(9):725-30. doi: 10.1093/ecco-jcc/jjv091. Epub 2015 May 19. PMID 25994356
- [Background] Borren NZ, van der Woude CJ, Ananthakrishnan AN. Fatigue in IBD: epidemiology, pathophysiology and management. Nat Rev Gastroenterol Hepatol. 2019 Apr;16(4):247-259. doi: 10.1038/s41575-018-0091-9. PMID 30531816
- [Background] Cohen BL, Zoega H, Shah SA, Leleiko N, Lidofsky S, Bright R, Flowers N, Law M, Moniz H, Merrick M, Sands BE. Fatigue is highly associated with poor health-related quality of life, disability and depression in newly-diagnosed patients with inflammatory bowel disease, independent of disease activity. Aliment Pharmacol Ther. 2014 Apr;39(8):811-22. doi: 10.1111/apt.12659. Epub 2014 Feb 20. PMID 24612278
- [Background] Jelsness-Jorgensen LP, Bernklev T, Henriksen M, Torp R, Moum BA. Chronic fatigue is associated with impaired health-related quality of life in inflammatory bowel disease. Aliment Pharmacol Ther. 2011 Jan;33(1):106-14. doi: 10.1111/j.1365-2036.2010.04498.x. Epub 2010 Oct 25. PMID 21083587
- [Background] Romberg-Camps MJ, Bol Y, Dagnelie PC, Hesselink-van de Kruijs MA, Kester AD, Engels LG, van Deursen C, Hameeteman WH, Pierik M, Wolters F, Russel MG, Stockbrugger RW. Fatigue and health-related quality of life in inflammatory bowel disease: results from a population-based study in the Netherlands: the IBD-South Limburg cohort. Inflamm Bowel Dis. 2010 Dec;16(12):2137-47. doi: 10.1002/ibd.21285. PMID 20848468
- [Background] van Gennep S, de Boer NKH, Gielen ME, Rietdijk ST, Gecse KB, Ponsioen CY, Duijvestein M, D'Haens GR, Lowenberg M, de Boer AGEM. Impaired Quality of Working Life in Inflammatory Bowel Disease Patients. Dig Dis Sci. 2021 Sep;66(9):2916-2924. doi: 10.1007/s10620-020-06647-y. Epub 2020 Oct 16. PMID 33063191
- [Background] Nocerino A, Nguyen A, Agrawal M, Mone A, Lakhani K, Swaminath A. Fatigue in Inflammatory Bowel Diseases: Etiologies and Management. Adv Ther. 2020 Jan;37(1):97-112. doi: 10.1007/s12325-019-01151-w. Epub 2019 Nov 23. PMID 31760611
- See also: Crohn's & Colitis Foundation. 2022. IBD and Fatigue. — https://www.crohnscolitisfoundation.org/pain-and-fatigue/fatigue-causes